CLINICAL TRIAL: NCT01359761
Title: Post Admission Cognitive Therapy (PACT) for the Inpatient Treatment of Military Personnel With Suicidal Behaviors: A Multi-Site Randomized Controlled Trial
Brief Title: Post Admission Cognitive Therapy (PACT) for the Inpatient Treatment of Military Personnel With Suicidal Behaviors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Duke University (Other); University of Michigan (Other); University of Pennsylvania (Other); Walter Reed National Military Medical Center (U.S. Federal Agency); Fort Belvoir Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marjan Holloway, Principal Investigator, Henry M. Jackson Foundation for the Advancement of Military Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-11-2-0106
Record Dates: First submitted 2011-05-17; First posted 2011-05-25 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Suicide, Attempted; Suicidal Ideation Active
Keywords: Suicide; Cognitive Therapy; Inpatient; Military
MeSH Terms: conditions — Suicide, Attempted; Suicide | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Post Admission Cognitive Therapy (PACT) (Experimental): Six (6) 60-90 Minutes Post Admission Cognitive Therapy Individual Sessions; Up to Two (2) Inpatient Booster Sessions; Up to Four (4) Telephone Booster Sessions Following Psychiatric Discharge; 12-Months Case Management
  Interventions: Behavioral: Post Admission Cognitive Therapy (PACT)
- Enhanced Usual Care (EUC) (No Intervention): Treatment As Usual and Study Assessment Services; 12-Months Case Management

INTERVENTIONS:
Behavioral: Post Admission Cognitive Therapy (PACT) — Six (60-90 minutes) individual psychotherapy sessions administered over preferably 3 days of inpatient stay, up to 2 booster sessions during hospitalization, and 4 telephone booster sessions within 3-months post discharge
  Other Names: Cognitive Therapy; Cognitive Behavior Therapy
  Arms: Post Admission Cognitive Therapy (PACT)

SUMMARY:
This study will implement and empirically evaluate the efficacy of a cognitive behavioral intervention program, titled, Post Admission Cognitive Therapy(PACT), for military service members and beneficiaries [with Veterans expected to be added] admitted for inpatient care due to severe suicide ideation and/or a recent suicide attempt.

DETAILED DESCRIPTION:
Background: Suicide remains a serious national public health problem and has become a leading cause of death in the United States military. To date, there is no evidence-based civilian or military inpatient interventions aimed at the reduction of suicide behavior. Our proposal addresses this important gap and aims to evaluate an innovative suicide intervention, Post Admission Cognitive Therapy (PACT). Left untreated, severe suicide ideation and/or suicide attempts that require psychiatric hospitalization may place an individual at a lifetime risk for increased psychopathology, subsequent suicide behavior, and death.

Objective: The broad objective is to implement and empirically evaluate the efficacy of a cognitive behavioral intervention program, titled Post Admission Cognitive Therapy (PACT), for military service members and beneficiaries [with Veterans expected to be added] admitted for inpatient care due to severe suicide ideation (with lifetime history of suicide attempt) and/or a recent suicide attempt.

Specific Aims: To evaluate the efficacy of PACT plus Enhanced Usual Care (EUC) versus EUC for the prevention of suicide in psychiatrically hospitalized military personnel and beneficiaries [with Veterans expected to be added] at follow-up (1, 3, 6, and 12-month) on (1) incidence of repeat suicide attempt(s) and number of days until a repeat suicide attempt (primary outcomes), and (2) psychiatric symptoms (depression, trauma, sleep, suicide ideation), repeat number of psychiatric hospitalization(s), hope for one's future, and acceptability of treatment (as measured by time to linkage to specialty care, attitudes toward seeking help for mental health issues, and subsequent mental health service utilization) (secondary outcomes). The investigators expect that adults in the PACT+EUC (experimental) condition compared to those in the EUC (control) condition will show favorable outcomes on both primary and secondary measures.

Study Design: The research design is a multi-site, single-blind, randomized controlled trial (RCT). A total of 218 individuals who are over the age of 18, able to communicate in English and willing to provide informed consent will be recruited from the inpatient psychiatric units at the Walter Reed National Military Medical Center and the Fort Belvoir Community Hospital [Washington DC VA expected to be added as third site]. Participants will be randomized into one of two conditions: (1) [Post Admission Cognitive Therapy (PACT) + Enhanced Usual Care (EUC)] or (2) Enhanced Usual Care (EUC). Individuals randomized into PACT+EUC will participate in the study assessments, receive six 60-90 minute individual face-to-face PACT psychotherapy sessions provided during their inpatient stay, up to a maximum of four 30-minute phone PACT booster sessions during the 3 months post hospital discharge, and case management services for 12 months. Individuals randomized into the control condition (EUC) will not receive the study intervention; they will receive the usual care provided in the inpatient setting, participate in study assessments, and receive case management services for 12 months. Patients in both conditions will be assessed on the dependent measures at baseline and at 1-, 3-, 6-, and 12-month follow-up intervals.

Relevance: Delivering a brief and possibly potent psychotherapeutic intervention during a psychiatric inpatient hospitalization followed by an aftercare component aims to directly target individuals at high risk for future suicide behavior, specifically psychiatrically hospitalized adults. The development and empirical validation of an inpatient cognitive behavioral treatment is a significant endeavor in our national as well as Department of Defense (DoD) suicide prevention efforts. If Post Admission Cognitive Therapy is found to be efficacious, the intervention can be subsequently disseminated to inpatient settings as the standard of care for military personnel and beneficiaries as well as Veterans admitted for suicide-related events.

ELIGIBILITY:
Inclusion Criteria:

* Reason for Admission: Suicide-Related Event
* Baseline Completed within Preferably 48-72 Hours of Admission
* Over the Age of 18
* Provides Informed Consent

Exclusion Criteria:

* Medical Incapacity to Participate
* Serious Cognitive Impairment
* Expected Discharge within 72 Hours of Admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2013-06-24 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Repeat Suicide Attempts | 1, 3, 6, and 12 months
  Repeat suicide attempts will be assessed using the Columbia Suicide Severity Rating Scale (C-SSRS) which documents the number of subsequent suicide attempts; medical records will also be checked.

SECONDARY OUTCOMES:
Depression | 1, 3, 6, and 12 months
  The Beck Depression Inventory-II (BDI-II) will be used to assess for symptoms of depression.
Hopelessness | 1, 3, 6, and 12 months
  The Beck Hopelessness Scale (BHS) will be used to assess for levels of hopelessness.
Suicide Ideation | 1, 3, 6, and 12 months
  The Scale for Suicide Ideation (SSI) and the Columbia Suicide Severity Rating Scale (C-SSRS) will be administered to assess for suicide-related thoughts (ideation), as well as the frequency, intensity, and specificity of these thoughts.
Post-Traumatic Stress Symptoms | 1, 3, 6, and 12 months
  The MINI Neuropsychiatric Interview and the PTSD Checklist (PCL) will be administered to assess for post-traumatic stress symptoms.
Acceptability of Treatment | 1, 3, 6, and 12 months
  Acceptability of treatment will be assessed by using Barriers to Care Items.
Repeat Psychiatric Hospitalizations | 1, 3, 6, and 12 months
  Subsequent psychiatric hospitalizations will be assessed for using the Cornell Services Index (CSI), as well as by accessing the Defense Medical Surveillance System (DMSS), which contains electronic medical records of all military personnel (permission to access participants' DMSS records is given at time of consent).

CONTACTS AND LOCATIONS:
Overall Officials: Marjan G Holloway, Ph.D., Principal Investigator — Uniformed Services University of the Health Sciences
Locations (4):
- United States (4):
  - Uniformed Services University of the Health Sciences, Bethesda, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Duke University, Durham, North Carolina
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghahramanlou-Holloway M, Neely L, Tucker J. A cognitive-behavioral strategy for preventing suicide. Current Psychiatry 13(8): 18-25, 2014.
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] LaCroix JM, Colborn VA, Hassen HO, Perera KU, Weaver J, Soumoff A, Novak LA, Ghahramanlou-Holloway M. Intimate partner relationship stress and suicidality in a psychiatrically hospitalized military sample. Compr Psychiatry. 2018 Jul;84:106-111. doi: 10.1016/j.comppsych.2018.04.006. Epub 2018 Apr 21. PMID 29747068